CLINICAL TRIAL: NCT03562689
Title: Cognitive Processing in Patients Surviving Delirium. Neuropsychological, EEG and Structural Brain Correlates.
Status: Suspended | Type: Observational
Why Stopped: Not enough subjects.
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Olalla Urdanibia Centelles, MD; PhD Candidate, Rigshospitalet, Denmark
Other Study IDs: 63657
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Septic Encephalopathy; Delirium; Sepsis
Keywords: Sepsis; Encephalopathy; Delirium; ICU; EEG; MRI; Cognitive tests
MeSH Terms: conditions — Sepsis-Associated Encephalopathy; Delirium; Sepsis; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Delirium and with septic encephalopathy. — Delirium or septic encephalopathy survivors will be analized in the same way: Cognitive tests, EEG and MRI.

SUMMARY:
The research program explores how delirium influenced brain function in patients surviving delirium and septic encephalopathy from a non neurological specialized ICU cohort from 2013 to 2015 in Rigshospitalet (Glostrup).

DETAILED DESCRIPTION:
The overall aim is to understand the pathophysiological mechanism in delirium and septic encephalopathy and its consequences.

For this purpose we will:

1. Provide extensive cognitive testing. These results provide the basis for categorization of patients surviving septic encephalopathy and delirious patients.
2. First, the investigators will examine if the differences in cognitive function is reflected in the ability of the brain to generate high-frequency electrical oscillations that accompany and underlie perception, attention, cognition, memory formation and retrieval. It will be performed by carrying out continuous EEG (cEEG) and by examination of steady-state evoked cognitive EEG responses.
3. Second, the investigations will examine MRI, structural and diffusion tensor imaging sequences. Hippocampal, thalamic, amygdala, lentiform nucleus and cingulate cortex volumes will be determined bilaterally and will be compared between individuals with healthy brain aging and patients that survived delirium.
4. Third, the investigators will assess plasma markers of free radical production.

ELIGIBILITY:
Inclusion Criteria for the ICU cohort:

* Age >18 years;
* Length of stay >24 hours in the ICU.

Exclusion Criteria for the ICU cohort:

* Expected death <24 hours;
* Psychiatric illness; pre-existing delirium; severe dementia; cerebrovascular event <six months; major surgery <two months;
* Non-Danish or English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Survivors of the critical ill cohort which were included the ones without known acute central nervous system affection admitted to a medical ICU with sepsis or septic shock, mono- or multi organ failure (respiratory insufficiency, circulatory shock, hepatic and/or renal failure) as indicated by a need for invasive or non-invasive mechanical ventilation, vasoactive drugs and/or CRR)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
EEG frequencies | Through study completion, an average of 1 year
  Automatically measurments of frequencies band
MRI | Through study completion, an average of 1 year
  Structural and diffusion tensor imaging sequences
Cognitive test: Verbal-Paired Associates | Through study completion, an average of 1 year
  Assessing explicit episodic memory performance
Cognitive test: Mini-Mental State Examination (MMSE) | Through study completion, an average of 1 year
  neurocognitive function
Cognitive test: Trail-Making Test and the Symbol-Digit Modalities Test (SDMT), | Through study completion, an average of 1 year
  Speed of processing and executive functioning

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
EEG, cognitive tests and MRI could be available for other researchers in the field.